CLINICAL TRIAL: NCT01360151
Title: Aqueous Humor Level of Cytokines in Polypoidal Choroidal Vasculopathy and Change of Cytokines After Photodynamic Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Ophthalmology, Professor, Seoul St. Mary's Hospital, Catholic University of Korea, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-Lee
Record Dates: First submitted 2011-04-12; First posted 2011-05-25 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-04

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: VEGF (Vascular endothelial growth factor)
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- experimental (Experimental): Arm 1 : combination treatment of ranibizumab(Lucentis) and verteporfin(Visudyne) injection
  Interventions: Drug: ranibizumab(Lucentis), verteporfin(Visudyne)
- active comparator (Active Comparator): Arm 2 : Treatment of verteporfin(Visudyne)
  Interventions: Drug: ranibizumab(Lucentis), verteporfin(Visudyne)
- normal control group (No Intervention): Arm 3 : normal control group
  Interventions: Drug: ranibizumab(Lucentis), verteporfin(Visudyne)

INTERVENTIONS:
Drug: ranibizumab(Lucentis), verteporfin(Visudyne) — ranibizumab(Lucentis) : 0.5mg/0.05ml - intravitreal injection verteporfin (Visudyne) : 15mg (6mg/m2)- intravenous injection
  Other Names: ranibizumab(Lucentis) : 0.5mg/0.05ml; verteportin (Visudyne) : 15mg (6mg/m2)

SUMMARY:
This is a prospective, comparative control analysis. The investigators want to evaluate the aqueous humor levels of vascular endothelial growth factor in polypoidal choroidal vasculopathy and the effect of photodynamic therapy and combination treatment of photodynamic therapy and Lucentis (Ranibizumab)on the level of vascular endothelial growth factor.

DETAILED DESCRIPTION:
To compare the effect of combination therapy of intravitreal injection of Lucentis™ and photodynamic therapy versus only photodynamic therapy on aqueous humor vascular endothelial growth factor level in polypoidal choroidal vasculopathy patients to establish the vascular endothelial growth factor expression after photodynamic therapy and the direct effect of Lucentis™ on this increased vascular endothelial growth factor level. Additionally the investigators want to examine the vascular endothelial growth factor , tumor necrosis factor alpha, interleukin-2, interleukin-6 and interleukin-8 level of aqueous humor in symptomatic, active polypoidal choroidal vasculopathy patients.

ELIGIBILITY:
<Polypoidal choroidal vasculopathy group>

Inclusion Criteria:

* Male or Female patients ≥ 45yrs of age
* Best corrected Visual acuity 20/30 to 20/320 Snellen equivalent using ETDRS chart measured at 4 meters
* Signed written informed consent
* Evidence of Polypoidal choroidal vasculopathy , active in disease activity.
* Presence of subfoveal, juxtafoveal or extrafoveal active characteristic macular polypoidal lesions on indocyanine green angiography
* Confirmed to be active in disease activity by fluorescein angiography
* The total lesion must have the greatest linear dimension less than 5400 microns ( ~9 MPS Disc Areas ) as delineated by indocyanine green angiography
* Had not been treated in the past
* Patients willing and able to comply with all study procedures

Exclusion Criteria:

* Previous history of laser photocoagulation,photodynamic therapy,anti VEGF therapy, submacular surgery in the study eye
* Have known hypersensitivity to Visudyne® and Lucentis™
* Previous treatment with external-beam radiation therapy or transpupillary thermotherapy
* History of vitrectomy
* Intraocular surgery,yttrium aluminum garnet(YAG) laser< 1month before day 0
* Additional eye disease that could compromise visual acuity
* Ocular inflammation
* Vitreous hemorrhage
* Uncontrolled glaucoma
* Current use or of likely need for systemic medications known to be toxic to the eye.
* Inability to obtain fluorescein angiography and indocyanine green angiography, due to media opacity, allergy to the dye or lack of venous access
* Are participating in another clinical study.
* Disciform scar
* Mental illness that precludes the patient from giving informed consent
* Patients who are considered potentially unreliable

<Control group>

-Age matched patients with cataract without other ocular diseases such as glaucoma, high myopia, ocular ischemic diseases, retinal disease, or with systemic diseases like diabetes mellitus.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
change from baseline in cytokine levels at 1 week, 1 month and 3 month | baseline, 1 week, 1 month, 3 month
  1. To compare the baseline level of cytokines in aqueous humor. polypoidal choroidal vasculopathy group(Arm A+Arm B) vs normal control group
  2. To compare the change of cytokine level of aqueous humor after combination treatment of intravitreal injection of Lucentis™ and photodynamic therapy versus only photodynamic therapy.(1 week, 1 month, 3 month)

CONTACTS AND LOCATIONS:
Locations (1):
- Won Ki Lee, Seoul, South Korea